CLINICAL TRIAL: NCT03483051
Title: Targeting Pulsatile Load to Increase Exercise Capacity and Quality of Life After Aortic Valve Replacement for Severe Aortic Stenosis (PULSE AS)
Acronym: PULSE-AS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 828994
Record Dates: First submitted 2018-02-15; First posted 2018-03-29 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic stenosis, aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — potassium nitrate; Potassium Chloride

STUDY DESIGN:
Intervention Model Description: In this phase IIb, double-blind, cross-over trial, we will assign 22 subjects who are post-TAVR for severe AS to: (A) Potassium nitrate administered by mouth at a dose of 6 mEq three times daily for 4 weeks, or (B) Potassium chloride (KCl) at identical doses. The order of the interventions (AB-BA design) will be randomized, with a 1-week washout period separating each intervention. A crossover design will enable each subject to receive both treatments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Potassium Nitrate (KNO3) (Experimental): Capsules containing 18 mmoles of KNO3 per day, given as one capsule (6 mmoles) three times a day for 4 weeks.
  Interventions: Drug: Potassium Nitrate
- Potassium Chloride (Sham Comparator): Capsules containing 18 mmoles of KCl per day, given as one capsule (6 mmoles) three times a day for 4 weeks.
  Interventions: Drug: Potassium Chloride

INTERVENTIONS:
Drug: Potassium Nitrate — Potassium nitrate capsules will consist of potassium nitrate (KNO3-) crystals [610 mg, corresponding to 6.03 mmoles of NO3-] with 190mg of lactose monohydrate, spray dried, NF. The dose for this trial will be 18 mmoles of NO3-per day, given as one capsule (6 mmoles) three times a day.
  Arms: Potassium Nitrate (KNO3)
Drug: Potassium Chloride — Potassium chloride capsules will consist of potassium chloride (KCl), granular, USP (450mg) plus lactose monohydrate, spray dried, NF (300mg). The dose for this trial will be 18 mmoles of KCl per day, given as one capsule (6 mmoles) three times a day.
  Arms: Potassium Chloride

SUMMARY:
The current trial is designed to assess the safety and efficacy of sustained oral administration of inorganic nitrate in patients with severe aortic stenosis and to assess the mechanisms by which inorganic nitrate enhances oxygen uptake and exercise capacity in this population.

DETAILED DESCRIPTION:
This is a randomized double-blind crossover clinical trial, in which 22 subjects who underwent transcatheter aortic valve replacement (TAVR) for severe aortic stenosis (AS) three or more months prior to enrollment will receive the following 2 interventions, in randomized order: (1) Potassium nitrate (KNO3), at a dose of 12-18 mmol/d by mouth for 4 weeks, or; (2) Potassium chloride (KCl), at a dose of 12-18 mmol/d by mouth for 4 weeks. A 1-week washout period will be introduced between the 2 interventions. The purpose of the trial is to test the safety of KNO3 and its efficacy on a number of clinical and physiologic endpoints in subjects who underwent TAVR for severe AS.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 50-90 years of age
2. Diagnosis of severe aortic stenosis prior to aortic valve repair
3. Successful trancatheter aortic valve repair via transfemoral procedural approach or successful surgical aortic valve repair at least three months prior to enrollment
4. Stable medical therapy: no addition/removal/changes in anti-hypertensive medications, or beta-blockers in the preceding 30 days.

Exclusion Criteria

1. Supine systolic blood pressure (SBP) < 100 mmHg OR supine diastolic blood pressure (DBP) <60 mmHg
2. Poorly controlled hypertension, as defined as SBP > 160 mmHg OR DBP > 100 mmHg
3. Pregnancy. Women of childbearing potential will undergo a pregnancy test during the screening visit
4. Atrial fibrillation within the prior 8 weeks before enrollment
5. Inability/unwillingness to exercise
6. Moderate or greater mitral regurgitation or aortic/peri-valvular regurgitation, any degree of mitral stenosis, severe right-sided valvular disease, or presence of a mitral prosthetic valve.
7. Moderate or severe patient prosthesis mismatch, as defined by Effective Orifice Area Index < 0.85 cm2/m2
8. Hypertrophic, infiltrative, or inflammatory cardiomyopathy
9. Pericardial disease
10. Current angina
11. Acute coronary syndrome or coronary intervention within the past 2 months
12. Primary pulmonary arteriopathy
13. Clinically significant lung disease as defined by: Chronic Obstructive pulmonary disease meeting Stage III or greater GOLD criteria, treatment with oral steroids within the past 6 months for an exacerbation of obstructive lung disease, or the use of daytime supplemental oxygen
14. Ischemia on stress testing without subsequent revascularization (during the screening visit)
15. Treatment with phosphodiesterase inhibitors that cannot be withheld
16. Treatment with organic nitrates
17. Significant liver disease impacting synthetic function or volume control (ALT/AST > 3x ULN, Albumin <3.0 g/dL)
18. eGFR < 30 mL/min/1.73 m2
19. G6PD deficiency. For males of African, Asian or Mediterranean decent, this will be evaluated prior to drug administration. A qualitative test positive for deficiency or a quantitative test with clinically significant G6PD deficiency (<60% of normal activity) will prompt exclusion from the trial (prior to drug administration).
20. History of methemoglobinemia or methemoglobin level >5% at baseline visit
21. Serum K>5.0 mEq/L
22. Severe right ventricular dysfunction.
23. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Chirinos, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject withdrew consent prior to treatment
  1 subject screen failed
Groups:
- ARM A Potassium Nitrate Then Potassium Chloride: Capsules containing 18 mmoles of KNO3 per day, given as one capsule (6 mmoles) three times a day for 4 weeks.
  Potassium Nitrate: Potassium nitrate capsules will consist of potassium nitrate (KNO3-) crystals [610 mg, corresponding to 6.03 mmoles of NO3-] with 190mg of lactose monohydrate, spray dried, NF. The dose for this trial will be 18 mmoles of NO3-per day, given as one capsule (6 mmoles) three times a day.
- ARM B Potassium Chloride Then Potassium Nitrate: Capsules containing 18 mmoles of KCl per day, given as one capsule (6 mmoles) three times a day for 4 weeks.
  Potassium Chloride: Potassium chloride capsules will consist of potassium chloride (KCl), granular, USP (450mg) plus lactose monohydrate, spray dried, NF (300mg). The dose for this trial will be 18 mmoles of KCl per day, given as one capsule (6 mmoles) three times a day.
Period: First Treatment, Pre Crossover
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Second Treatment, After Crossover
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 subject withdrew consent prior to enrollment
  1 subject was a screen failure and never received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Work Performed During a Maximal-effort Exercise Test
Description: The effect of KNO3 on exercise capacity, quantified as Total work performed during a maximal-effort exercise test;
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Peak Oxygen Uptake (VO2) During a Maximal Effort Exercise Test
Description: The effect of KNO3 on exercise capacity, quantified as: Peak oxygen consumption (VO2) during a symptom-limited maximal effort exercise test.
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Quality of Life Score
Description: The effect of KNO3 on quality of life, assessed using the Kansas City Cardiomyopathy Questionnaire.
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Systemic Vasodilator Response to Exercise
Description: The effect of KNO3 on systemic vasodilator response, measured by change in systemic vascular resistance, during a symptom-limited maximal exercise test,
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Left Ventricle Diastolic Function
Description: The effect of KNO3 on left ventricle diastolic filling parameters (measured with echocardiography at rest and after peak exercise)
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Myocardial Systolic Strain
Description: The effect of KNO3 on myocardial strain (assessed with speckle-tracking echocardiography)
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Late Systolic Left Ventricle Load
Description: The effect of KNO3 on last systolic left ventricle load from wave reflections (assessed via comprehensive aortic pressure-flow regulations, using arterial tonometry and Doppler echocardiography)
Time Frame: 9 weeks
Population: Efficacy data analyses cannot be reported for privacy reasons due to enrollment of only three (3) subjects.
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | ARM A Potassium Nitrate Then Potassium Chloride | ARM B Potassium Chloride Then Potassium Nitrate
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A Potassium Nitrate Then Potassium Chloride (N=2) | ARM B Potassium Chloride Then Potassium Nitrate (N=1)
Lightheadedness (Cardiac disorders) | 2 (2) | 0 (0)
Stomach Ache, diarrhea, nausea or vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drop in blood pressure when standing up (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Efficacy data analyses will not be performed as they are not meaningful due to enrollment of only three (3) subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03483051/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03483051/ICF_001.pdf